CLINICAL TRIAL: NCT01951469
Title: Multicenter Phase III Study of Gefitinib Mono-therapy or Gefitinib Combined With Chemotherapy in Patients With Brain Metastases From Non-small Cell Lung Cancer Harboring EGFR Mutation
Brief Title: Gefitinib With or Without Chemotherapy in Brain Metastases From Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Wu Jieping Medical Foundation (Other)
Responsible Party: Principal Investigator, Li-kun Chen, medical doctor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSCLC brain metastasis 01
Record Dates: First submitted 2013-09-16; First posted 2013-09-26 (Estimated); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Non-small Cell Lung Cancer; Brain Metastases; EGFR Mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — Gefitinib; Pemetrexed; Platinum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gefitinib and Pemetrexed/platinum (Experimental): Gefitinib 250mg is Taken Orally on day 1-28,combined Pemetrexed (D1)+cisplatin (D1-3) chemotherapy or Pemetrexed (D1)+nedaplatin (D1) chemotherapy, every 28 days
  Interventions: Drug: Gefitinib and Pemetrexed/platinum
- Gefitinib mono-therapy (Active Comparator): Gefitinib 250mg is Taken Orally everyday
  Interventions: Drug: Gefitinib mono-therapy

INTERVENTIONS:
Drug: Gefitinib and Pemetrexed/platinum — Gefitinib 250mg is Taken Orally on day 1-28,combined Pemetrexed (D1)+cisplatin (D1-3) or Pemetrexed (D1) + nedaplatin (D1) chemotherapy, every 28 days
  Arms: Gefitinib and Pemetrexed/platinum
Drug: Gefitinib mono-therapy — Gefitinib 250mg is Taken Orally everyday
  Arms: Gefitinib mono-therapy

SUMMARY:
This is a multi-center phase III randomized controlled study to assess the efficacy of Gefitinib alone and Gefitinib combination with Pemetrexed/platinum on patients with brain metastasis from non-small cell lung cancer(NSCLC) harboring EGFR mutation type by intracranial PFS(iPFS),also PFS ,DCR and OS.The side effect is evaluated as well.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who was confirmed stage IV NSCLC with EGFR activating mutation and brain metastases by pathologic histology or cytology
2. Patients who had never received therapy (including chemotherapy,WBRT,EGFR-TKI and EGFR monoclonal antibody) after diagnosed brain metastases
3. Patients had at least three metastatic lesions in brain, or patients with 1-2 intracranial lesions who were not suitable for brain radiotherapy, or patients with 1-2 intracranial lesions who refused brain radiotherapy, at least one intracranial lesion with the longest diameter of >5 mm
4. Adult patients (≥ 18 years and ≤75 years). ECOG Performance Status 0 or 1 Life expectancy of at least 12 weeks.,Haemoglobin ³ 10.0 g/dl, Absolute neutrophil count (ANC) ³1.5 x 109/L, platelets ³ 100 x 109/L. Total bilirubin £ 1.5 x upper limit of normal (ULN). ALT and AST < 2.5 x ULN in the absence of liver metastases, or < 5 x ULN in case of liver metastases. Creatinine clearance ³ 60ml/min (calculated according to Cockcroft-gault formula).
5. Patients should be contraceptive during the period of the trial until 8 weeks after the last administration of icotinib.
6. Able to comply with the required protocol and follow-up procedures, and able to receive oral medications.

Exclusion Criteria:

1. Patient was received irradiation of brain. Patient with meningeal metastases were confirmed by MRI or cytology test of cerebrospinal fluid.
2. Patient is received the treatment of Phenytoin, carbamazepine, rifampicin, phenobarbital, or St. John's Wort.
3. Patient was received EGFR Tyrosine Kinase Inhibitor or EGFR monoclonal antibody.
4. Interstitial pneumonia.Pericardial effusion, pleural effusion is uncontrolled .
5. Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease).
6. Any significant ophthalmologic abnormality ,especially severe dry eye syndrome ,keratoconjunctivitis sicca,Sjogren syndrome,severe exposure keratitis or any other disorder likely to increase the risk of corneal epithelial lesions.
7. Lack of physical integrity of the upper gastrointestinal tract, or malabsorption syndrome, or inability to take oral medication, or have active peptic ulcer disease.
8. The symptoms of increased intracranial pressure are uncontrolled after dehydration and cortisone treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
iPFS(intracranial progression free survival | 2 years
  defined as time from randomization to intracranial progressive disease or death.

SECONDARY OUTCOMES:
ORR | 2 years
  proportion of patients with complete or partial response of overall lesions
intracranial objective response rate (iORR) | 2 years
  proportion of patients with complete or partial response of intracranial lesions
PFS(Progression Free Survival) | 2 years
  time from randomization to overall disease progression or death
OS(Overall Survival) | 3 years
  time from randomization to death from any cause
adverse events | 3 years
  adverse events were evaluated according to NCI-CTCAE 4.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University of Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Hou X, Li M, Wu G, Feng W, Su J, Jiang H, Jiang G, Chen J, Zhang B, You Z, Liu Q, Chen L. Gefitinib Plus Chemotherapy vs Gefitinib Alone in Untreated EGFR-Mutant Non-Small Cell Lung Cancer in Patients With Brain Metastases: The GAP BRAIN Open-Label, Randomized, Multicenter, Phase 3 Study. JAMA Netw Open. 2023 Feb 1;6(2):e2255050. doi: 10.1001/jamanetworkopen.2022.55050. PMID 36753281